CLINICAL TRIAL: NCT05467514
Title: Effect of Liraglutide on Subclinical Atherosclerosis in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: David Sanchez Garcia (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor-Investigator, David Sanchez Garcia, Principal Investigator David Sanchez Garcia, Instituto Mexicano del Seguro Social
Organization: Instituto Mexicano del Seguro Social (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F-2022-1901-019
Record Dates: First submitted 2022-07-07; First posted 2022-07-20 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Liraglutide; Diabetes Mellitus, Type 1; Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Atherosclerosis | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: Application of liraglutide 1.8 mg subcutaneous daily for 6 months to evaluate subclinical atherosclerosis, by means of carotid doppler US, lipid profile in patients with type 1 diabetes mellitus
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liraglutide (Experimental): Application of liraglutide 1.8 mg subcutaneous daily for 6 months to evaluate subclinical atherosclerosis, by means of carotid doppler US, lipid profile in patients with type 1 diabetes mellitus
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Application of liraglutide 1.8 mg subcutaneous daily for 6 months to evaluate subclinical atherosclerosis, by means of carotid doppler US, lipid profile in patients with type 1 diabetes mellitus

SUMMARY:
The aim of the trail is investigate the effect of liraglutide 1.8mg as add-on to insulin for 6 months on carotid intima media thickness and cardiovascular risk factors in subjects with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Age from 15 to 60 years
* Patients diagnosed with Type 1 Diabetes Mellitus.
* Diabetes duration more than 1 year.
* Both genders.
* C - peptide less than 0.3 nmol/L

Exclusion Criteria:

* Patients with type 2 diabetes mellitus, LADA (latent autoimmune diabetes in adults), MODY (maturity-onset diabetes of youth), or other types of diabetes other than type 1 diabetes mellitus.
* Pregnant patients or desire to become pregnant in the next 6 months.
* Family history of medullary thyroid cancer or multiple endocrine neoplasia 2
* History of pancreatitis
* Familial hypercholesterolemia
* Use of adjunctive treatment to insulin (SGLT-2 [sodium-glucose cotransporter-2] inhibitor, Pramlintide, metformin)
* Start of treatment with statins, ezetimibe or PSCK9 (proprotein convertase subtilisin/kexin type 9) inhibitors, amlodipine, metoprolol in the last 6 months before the study.
* Bariatric surgery
* Use of medications (immunosuppressants, calcineurin inhibitors, mTOR (mammilian target of rapamycin) inhibitors, corticosteroids, aspirin, or anticoagulants)
* Metabolic abnormalities (inborn errors of cholesterol storage metabolism, glycogen storage, abetalipoproteinemia, Reye's disease, LCAT (lecithin-cholesterol acyltransferase) deficiency)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
To assess the effect of liraglutide on carotid intima media thickness in patients with type 1 diabetes mellitus. | Baseline and 6 months
  Change from baseline measure of right carotid intima media thickness with doppler ultrasound at 6 months in patients with type 1 diabetes mellitus who meet inclusion criteria.

SECONDARY OUTCOMES:
To assess the effect of liraglutide on cardiovascular risk factors, cardiometabolic markers (BMI, weight and abdominal circumference) | 0, 1, 2, 3, 4, 5 and 6 months
  Somatometry: weight will be measured at baseline and every month until completing 6 months.
To assess the effect of liraglutide on cardiovascular risk factors, cardiometabolic markers. Somatometry (BMI, weight and abdominal circumference) | 0, 1, 2, 3, 4, 5 and 6 months
  Somatometry: Body mass index will be measured at baseline and every month until completing 6 months.
To assess the effect of liraglutide on cardiovascular risk factors, cardiometabolic markers. Somatometry (BMI, weight and abdominal circumference) | 0, 1, 2, 3, 4, 5 and 6 months
  Somatometry: abdominal circumference will be measured at baseline and every month until completing 6 months.
To assess the effect of liraglutide on cardiovascular risk factors, cardiometabolic markers Laboratory studies (total cholesterol, LDL, HDL, triglycerides, non-HDL cholesterol) | 0, 3 and 6 months
  Laboratory studies will be taken: complete lipid profile (total cholesterol, LDL, HDL, triglycerides, non-HDL cholesterol) at baseline, 3 and 6 months.
To assess the effect of liraglutide on cardiovascular risk factors, cardiometabolic markers Laboratory studies (HbA1c) | 0, 3 and 6 months
  Laboratory studies will be taken: HbA1c at baseline, 3 and 6 months.
To assess the effect of liraglutide on cardiovascular risk factors, cardiometabolic markers. eGDR (Estimated glucose disposal rate) | 0, 3 and 6 months
  Estimated glucose disposal rate will be calculated at baseline, 3 and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Nacional del Noreste Hospital de Especialidades UMAE 25, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided